CLINICAL TRIAL: NCT05210166
Title: Transcutaneous Spinal Cord Stimulation Combined With Robot-assisted Therapy in Incomplete Spinal Cord Injury Patients.
Brief Title: Transcutaneous Spinal Cord Stimulation and Robotic Therapy
Acronym: tscs_Lokomat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Fundacion del Hospital Nacional de Paraplejicos para la Investigacion y la Integracion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ExoStim Project
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries
Keywords: Neuromodulation; Spinal cord injury; Robotics; Transcutaneous spinal cord stimulation; Lokomat
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: It is a double-blind, randomized, controlled clinical trial.
  There will be two groups:
  Group A (n=15): tSCS combined with Lokomat Group B (n=15): Sham-tSCS combined with Lokomat
Who Masked: Participant, Outcomes Assessor
Masking Description: For blinding of participants:
  The protocol will be the same in the active tSCS and sham tSCS groups. The sham stimulation will consist of the same stimulation parameters used for active tSCS, except for the stimulus intensity, which will be set at the sensory threshold, maintained for 30 s and then slowly decreased to zero. The participants will receive the same instructions that given to the active tSCS session.
  For blinding of outcomes assessor:
  Two blinded assessors will perform the evaluations before, after and a follow-up at 4 weeks post-intervention.
  The operator of the Lokomat will be also masked to the group allocation. To ensure this, the same stimulator and electrode location will be used for both groups and the screen of the device will be covered. Only the investigator who applies spinal stimulation will know which group belongs the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tSCS and Lokomat (Active Comparator): 20 sessions, 5 sessions per week of active transcutaneous spinal cord stimulation (tSCS) combined with Lokomat will be performed.
  The duration of Lokomat will be 30 minutes, of which the first 20 minutes tSCS will be applied at the beginning of each session.
  Interventions: Device: Active tSCS and Lokomat
- Sham tSCS and Lokomat (Placebo Comparator): 20 sessions, 5 sessions per week of sham transcutaneous spinal cord stimulation (sham-tSCS) combined with Lokomat will be performed.
  The duration of Lokomat will be 30 minutes, of which the first 20 minutes sham-tSCS will be applied at the beginning of each session.
  Interventions: Device: Sham tSCS and Lokomat

INTERVENTIONS:
Device: Active tSCS and Lokomat — A symmetrical biphasic 30 Hz current of 1 ms pulse-width with an electro-stimulator will be applied.
  For the stimulation intensity, the maximum intensity tolerated by the patient will be selected. The intensity will be increased in case of habituation to the current.
  Other Names: Experimental
  Arms: Active tSCS and Lokomat
Device: Sham tSCS and Lokomat — The protocol and device of sham tSCS combined with Lokomat will be the same as active tSCS except for the stimulus intensity, which will be set at the sensory threshold, maintained for 30 seconds and then slowly will be decreased to zero, being this intensity maintained for the remaining 20 minutes of stimulation.
  Other Names: Controlled
  Arms: Sham tSCS and Lokomat

SUMMARY:
Lumbosacral spinal stimulation activates the neural network involved in the control of locomotion at the spinal level. However, its effects are limited to the production of robust rhythmic patterns of alternating movement, being currently in the absence of therapeutic value. On the other hand, the use of robotic technology for gait rehabilitation has experienced significant growth during the last years and its clinical efficacy is similar to others traditional interventions.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) often results in complete or partial paralysis below the level of lesion, having a profound physical, psychological and socioeconomic impact on the affected person's life. Between the different approaches for the rehabilitation of SCI, we can find robot therapy. Robot-assisted gait training has emerged as a promising therapy for improving walking ability, balance and motor function in neurological patients. The underlying principle of this therapy is based on the execution of repetitive and task-specific training able to generate appropriate afferent inputs, activating the central pattern generators in the lumbosacral spinal cord. Another novel therapy is the use of transcutaneous spinal cord stimulation (tSCS), applied through self-adhesive electrodes in the skin. tSCS activates similar mechanisms than epidural stimulation and is able to stimulate the spinal locomotor circuits in SCI patients. It allows the activation of rhythmic, flexo-extension movements in the paralyzed lower limbs.

The aim of this study is to analyze the feasibility, safety and efectiveness of a program of 20 sessions of 30 Hz-tSCS applied over T11-12 intervertebral space combined with Lokomat training in patients with incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

* AIS C or D.
* 2-6 months after injury.
* Neurological level of injury between C4-T11.
* Ashworth less or equal 2.
* Penn less or equal 2.
* To understand and to sign the informed consent.

Exclusion Criteria:

* Metal implants over T11-T12
* Electronic device implants.
* Epilepsy
* Allergy to the electrode material
* Pregnancy
* Concomitant pathologies
* Pathology or fracture of the lower limbs
* Musculoskeletal injury in the lower limbs
* Lower limbs dysmetria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Change in isometric maximal voluntary contraction strength | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Isometric Maximal Voluntary Contraction Strength of quadriceps and tibialis anterior will be measured by hand-held dynamometer Micro Fet 2TM (Hoggan Scientific, LLC, Utah, USA) and will be expressed in Kgs.
Change in lower limbs muscle strength (LEMS) | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Lower limb muscle strength will be measured by Lower Extremity Motor Score (LEMS). The scores vary from 0-5 for each of five key muscles of the right and left lower limbs, with a maximum score of 50 for both lower extremities.

SECONDARY OUTCOMES:
Change in lower limbs spasticity | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Spasticity will be measured by the modified Ashworth scale (MAS). Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.
Change in peak-to-peak amplitude and latency of motor evoked potentials | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Motor evoked potentials (MEP) will be elicited by transcranial magnetic stimulation (TMS, Magstim Rapid) using a double-cone coil. The optimal stimulation site will be identified for the anterior rectus and tibialis anterior muscles individually with reference to the standard CZ point.
  MEP threshold will be defined as the minimal TMS intensity required to evoke a motor response (>0.1 mV peak-to-peak amplitude) during slight tonic contraction of the target muscle (approximately 20% of the isometric MVC). Test MEPs during the protocol will be recorded during 20% MVC as an average of in response to 10 single-pulse stimuli that will be applied at 120% of the MEP threshold.
Change in gait function | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  10-meter walk test (10MWT) will be expressed in seconds.
Change in balance and fall risk | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Test timed up and go (TUG) will be expressed in seconds. ≥12 seconds to complete the TUG means a higher risk for falling.
Change in aerobic capacity and endurance | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  The six-minute walk test will be expressed in meters. An increase in the distance walked indicates improvement in basic mobility.
Change in walking ability | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  Walking Index for Spinal Cord Injury (WISCI-II) assess the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from Spinal Cord Injury (SCI).
Change in daily function | Baseline, post-treatment (after 20 sessions) and follow-up at 4 weeks.
  The Spinal Cord Independence Measure (SCIM-III) is a scale for the assessment of achievements of the daily function of patients with spinal cord injury (SCI). The third version (SCIM III) contains 19 tasks organized in 3 subscales: self-care, respiration and sphincter management, and mobility. Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence.
Blinding assesment | At follow-up at 4 weeks.
  The success of participant and assessor blinding will be evaluated through a questionnaire after each intervention (active-tSCS and sham-tSCS) with five questions:
  (1) "Strongly believe the applied intervention is new treatment"; (2) "Somewhat believe the applied intervention is new treatment"; (3) "Somewhat believe the applied intervention is a placebo", (4) "Strongly believe the applied intervention is a placebo", or (5) "Do not know".

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gómez-Soriano, PhD, Study Director — Castilla La Mancha University
Locations (1):
- Castilla-La Mancha University, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comino-Suarez N, Moreno JC, Megia-Garcia A, Del-Ama AJ, Serrano-Munoz D, Avendano-Coy J, Gil-Agudo A, Alcobendas-Maestro M, Lopez-Lopez E, Gomez-Soriano J. Transcutaneous spinal cord stimulation combined with robotic-assisted body weight-supported treadmill training enhances motor score and gait recovery in incomplete spinal cord injury: a double-blind randomized controlled clinical trial. J Neuroeng Rehabil. 2025 Jan 30;22(1):15. doi: 10.1186/s12984-025-01545-8. PMID 39885542